CLINICAL TRIAL: NCT01962558
Title: A Blinded Randomized Pilot Study Assessing Vagus Nerve Stimulation (VNS) Paired With Tones for Tinnitus vs. VNS With Unpaired Tones
Brief Title: Vagus Nerve Stimulation (VNS) Paired With Tones for Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MicroTransponder Inc. (Industry)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MT-T-02; 2U44DC010084-04 (NIH)
Record Dates: First submitted 2013-10-09; First posted 2013-10-14 (Estimated); Results first posted 2018-04-06 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-03

CONDITIONS: Tinnitus
Keywords: Tinnitus; Medical Device; Randomized; Vagus Nerve Stimulation
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VNS Treatment (Experimental): Vagus nerve stimulation and tones are used 2.5 hours per day for a 6-week period.
  Interventions: Device: VNS Treatment
- VNS Control (Sham Comparator): Vagus nerve stimulation and tones are given daily over a 2.5 hour period, but not in the same way as the experimental group, and in such a way that it is believed to be ineffective but still provide both VNS and tones so that blinding is maintained.
  Interventions: Device: VNS Control

INTERVENTIONS:
Device: VNS Treatment — VNS is given in brief bursts over a 2.5 hour period. The subject also has headphone connected to a computer, and hears audio tones through the headphones that occur during VNS.
  Other Names: VNS paired with tones; Serenity System
  Arms: VNS Treatment
Device: VNS Control — This is the sham-control group; subjects in this group will receive both tones and VNS, but in a manner that is expected to be ineffective.
  Arms: VNS Control

SUMMARY:
Assess the safety and efficacy of VNS paired with tones for tinnitus using a randomized, controlled, parallel study design.

DETAILED DESCRIPTION:
Patients who have moderate to severe tinnitus, at least one year post diagnosis, may enroll. All patients will be implanted and randomized to one of two groups:

* a group receiving VNS paired with tones and;
* a group that receives VNS and tones, but with different settings.

After device use training, therapy is delivered at home by the patient for 6 weeks. Patients have eight baseline audiometric assessments along with two questionnaire assessments, an assessment after recovery before treatment starts, and tinnitus assessments every two weeks during therapy through the 6 week randomized portion of the study. After the randomized portion, all patients receive VNS paired with tones. Patients will continue to return for quarterly visits and tinnitus assessments through the first year after implant, regardless of their therapy status. Interested patients can continue to receive longer-term treatment after the first year. A goal of up to 30 patients enrolled and implanted across four sites is planned for this study.

ELIGIBILITY:
Inclusion Criteria:

1. 22 to 65 years of age
2. Have been diagnosed as suffering from sensorineural tinnitus and at least some tonal quality of the tinnitus
3. Unilateral or bilateral tinnitus
4. Have experienced tinnitus for at least one year and failed at least one tinnitus therapy (such as a counseling or sound therapy procedure. The diagnosis of tinnitus will include an audiological or medical diagnosis in their health records, as well as a patient affirmation of tinnitus greater than 12 months
5. MML >= 7 dB (decibel)
6. Have tinnitus score of 40 or greater on the Tinnitus Handicap Questionnaire; (THQ)
7. No tinnitus treatment for at least 4 weeks prior to study entry.
8. Willing and able to understand and comply with all study-related procedures during the course of the study

Exclusion Criteria:

1. Acute or intermittent tinnitus
2. Severe hearing loss in any ear, as defined as more than an 80 dB HL (decibels hearing level) at frequencies from 250 Hz. to 8,000 Hz.
3. Meniere's disease, ear tumors, or evidence of active middle ear disease (such as fluid, infection, tumor, mass)
4. Any other implanted device such as a pacemaker or other neurostimulator; any other investigational device or drug
5. Pregnant or plan on becoming pregnant or breastfeeding during the study period
6. Currently require, or likely to require, MRI or diathermy during the study duration
7. History of adverse reactions to anesthetics (e.g., lidocaine) that in the Investigator's opinion make surgery too risky
8. Beck Depression Inventory (BDI) of 30 or greater
9. Any other form of tinnitus treatments (e.g. Herbal medication, acupuncture or chiropractic medicine) are not allowed during the study.
10. Any drug known to mimic, increase or decrease release or removal of a diffuse neuromodulator, such as norepinephrine, dopamine, serotonin, benzodiazepines, and acetylcholine is not allowed, as well as any psychoactive medications.
11. Significant cardiac history
12. Use of any medication known to cause or increase tinnitus, such as NSAIDS (ibuprofen, naproxen, nabumetone, etc.), aspirin and other salicylates, furosemide (Lasix) and other "loop" diuretics, "mycin" antibiotics such as vancomycin, quinine and related drugs, and chemotherapy agents such as cisplatin.
13. Involvement in litigation (e.g., worker's compensation claim and/or receiving disability benefits related to tinnitus and/or hearing loss).

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-02; Primary Completion 2015-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W Brent Tarver, BSEE, Study Director — MicroTransponder Inc.
Locations (3):
- United States (3):
  - U. Iowa, Iowa City, Iowa
  - U. Buffalo, Buffalo, New York
  - UT Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) is not planned to be shared.

REFERENCES:
- [Background] Engineer ND, Moller AR, Kilgard MP. Directing neural plasticity to understand and treat tinnitus. Hear Res. 2013 Jan;295:58-66. doi: 10.1016/j.heares.2012.10.001. Epub 2012 Oct 23. PMID 23099209
- [Background] Engineer ND, Riley JR, Seale JD, Vrana WA, Shetake JA, Sudanagunta SP, Borland MS, Kilgard MP. Reversing pathological neural activity using targeted plasticity. Nature. 2011 Feb 3;470(7332):101-4. doi: 10.1038/nature09656. Epub 2011 Jan 12. PMID 21228773
- [Background] Tyler R, Cacace A, Stocking C, Tarver B, Engineer N, Martin J, Deshpande A, Stecker N, Pereira M, Kilgard M, Burress C, Pierce D, Rennaker R, Vanneste S. Vagus Nerve Stimulation Paired with Tones for the Treatment of Tinnitus: A Prospective Randomized Double-blind Controlled Pilot Study in Humans. Sci Rep. 2017 Sep 20;7(1):11960. doi: 10.1038/s41598-017-12178-w. PMID 28931943
- See also: Link to study website — http://www.tinnitustrial.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty-two subjects were screened for inclusion into the study. Nine (9) did not meet inclusion criteria, 15 declined to participate, 3 had medical issues, and 5 were screened but were after the study limit of 30. Thirty subjects were enrolled and implanted with the study device.
Period: Overall Study
Arm/Group | VNS Treatment | VNS Control
Started | 16 | 14
Acute Study | 16 | 14
12-Weeks | 16 | 14
Completed | 16 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with tinnitus
Groups:
- Total: Total of all reporting groups
Arm/Group | VNS Treatment | VNS Control | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (7.6) | 54.9 (9.1) | 55.6 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 10 | 11
  Male | 15 | 4 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 14 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events
Description: Assess the number of serious adverse events during the study, and compare between groups to indicate if there are more in the treatment group than the control group.
Time Frame: 6-weeks
Measure: Number; unit: participants
Arm/Group | VNS Treatment | VNS Control
Number analyzed (Participants) | 16 | 14
participants | 1 | 2

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Assess the number of adverse events during the study, and compare between groups to indicate if there are more in the treatment group than the control group.
Time Frame: 6-weeks
Measure: Number; unit: participants
Arm/Group | VNS Treatment | VNS Control
Number analyzed (Participants) | 16 | 14
participants | 11 | 9

3. Secondary Outcome: Change in Minimum Masking Level (MML) in Units of dB (Decibels)
Description: Asses the change in minimum masking level (MML) for both groups and compare between the groups.
Time Frame: 6-weeks (pre-implant to after 6-weeks of VNS)
Measure: Mean (95% Confidence Interval); unit: dB (decibels)
Arm/Group | VNS Treatment | VNS Control
Number analyzed (Participants) | 16 | 14
dB (decibels) | 3.5 [-.4 to 7.5] | -3.8 [-11.9 to 4.1]

4. Secondary Outcome: Percent Change in Tinnitus Handicap Inventory (THI)
Description: Assess the change in THI score for both groups and compare between the groups. The THI is a questionnaire that asks subjects to assess their perception of their tinnitus by rating each question as a Yes (4 points), No (0 points) or Sometimes (2 points). There are 25 questions, scores are summed, so the scale ranges from 0 to 100. Scores are graded as: Grade 1 - Slight (0-16) Only heard in a quiet environment; Grade 2 - Mild (18-36) Easily masked by environmental sounds and easily forgotten with activities.; Grade 3 - Moderate (38-56) Noticed in presence of background noise, although daily activities can still be performed.; Grade 4 - Severe (58-76) Almost always heard, leads to disturbed sleep patterns and can interfere with daily activities.; Grade 5 - Catastrophic (78-100) Always heard, disturbed sleep patterns, difficulty with any activities.
Time Frame: 6-weeks (pre-implant to after 6-weeks of VNS)
Measure: Mean (95% Confidence Interval); unit: percentage change of THI
Arm/Group | VNS Treatment | VNS Control
Number analyzed (Participants) | 16 | 14
percentage change of THI | -17.7 [-28 to -7.3] | -7.3 [-27.5 to 12.7]

5. Secondary Outcome: Change in Tinnitus Handicap Questionnaire (THQ)
Description: Assess the change in THQ score for both groups and compare between the groups. The THQ is a patient questionnaire with 27 questions with each question having a score from 1 to 100. Scoring includes three factors - Factor 1 (Social, Emotional, Behavioral), Factor 2 (Tinnitus and Hearing), Factor 3 (Outlook). Fifteen questions are included in Factor 1, 8 questions in Factor 2, and 4 questions in Factor 3. A total score is calculated by adding the scores for Factor 1 questions and multiplying by 15/27, adding the scores for Factor 2 and multiplying by 8/27, and adding the scores for Factor 3 and multiplying by 4/27. This is then summed for the total score. Total score ranges from 0 to 100, with higher scores indicating more severe tinnitus.
Time Frame: 6-weeks (pre-implant to after 6-weeks of VNS)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | VNS Treatment | VNS Control
Number analyzed (Participants) | 16 | 14
units on a scale | -2.5 [-8.3 to 3.3] | -7.5 [-15.8 to .7]

6. Other Pre Specified Outcome: Change in Tinnitus Functional Index (TFI)
Description: Assess the change in TFI score for both groups and compare between the groups. The TFI has eight subscales that address the intrusiveness of tinnitus, the sense of control the patient has, cognitive interference, sleep disturbance, auditory issues, relaxation issues, quality of life, and emotional distress. There are a total of 25 questions, with a range of 0 to 10 on each item (0 to 250) total. All valid answers are summed, divided by the number of questions which were answered, and multiplied by 10 (0-100 range). Score range from 0 to 100 with higher scores indicating worse tinnitus.
Time Frame: 6-weeks (pre-implant to after 6-weeks of VNS)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | VNS Treatment | VNS Control
Number analyzed (Participants) | 16 | 14
units on a scale | -2.03 [-7.1 to 3.1] | -7.5 [-15.5 to 0.7]

ADVERSE EVENTS:
Arm/Group | VNS Treatment | VNS Control
Serious Adverse Events (participants affected / at risk) | 1/16 | 2/14
Other Adverse Events (participants affected / at risk) | 2/16 | 1/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VNS Treatment (N=16) | VNS Control (N=14)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — Hoarseness due to damage to the vagus nerve; recovers over time.
Surgery (Surgical and medical procedures) | 0 (0) | 1 (1) — Surgery to replace broken lead
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VNS Treatment (N=16) | VNS Control (N=14)
Coughing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No